CLINICAL TRIAL: NCT05204680
Title: Exercise in Advanced Parkinson's Disease (PD) With Deep Brain Stimulation (DBS)
Acronym: DBS Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-500-203-70-04
Record Dates: First submitted 2021-12-23; First posted 2022-01-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic Exercise (Experimental): The participant will work with the physical therapist on an exercise regimen and first session will be supervised with the therapist. Exercise protocols will include a 15-minute warmup and cooldown session as well. To allow for increased participation and accessibility, the means of aerobic exercise will not be restricted and any safe mechanism of exercise will be allowed e.g., treadmill, stationary bike, etc.
  Subjects will be provided an activity monitor (Phillips HealthBand Monitor) for the duration of study participation and receive training on how to use it, including marking events with start and stop of exercise sessions and tracking heart rate. The device can track type of activity as well as cardio fitness index and VO2max.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — The participant will work with the physical therapist on an exercise regimen.

SUMMARY:
This project is a 3-month prospective study assessing the immediate and long-term changes associated with aerobic exercise in quality-of-life measures, nonmotor scores, brief neuropsychological batteries, and local field potentials (LFPs) in those with Parkinson's Disease (PD) who have undergone deep brain stimulation (DBS) surgery for management of their symptoms. In this study, the investigators will assess the feasibility of an aerobic exercise regimen in those with advanced PD and DBS, characterize the immediate and long-term changes in neuronal activity with exercise in PD, and assess the nonmotor impact of exercise in individuals with advanced PD and DBS.

The investigators will recruit individuals who are not regular exercisers and develop an individualized 3-month exercise plan with the assistance of physical therapists, using heart rate targets for moderate exercise. Outcomes will be measured at baseline and following 3-months of regular exercise. Field potentials will be noted at baseline, during exercise every 2 weeks, and then a final baseline at the end of 3 months in on-medication and on-stimulation states. This will allow for characterization of field potential changes over time both during exercise as efficiency improves as well as impact on baseline neuronal activity in the resting state. This study is novel in that most aerobic exercise studies target early PD subjects and rarely include those who have undergone DBS surgery. The study will specifically focus on the feasibility of developing an aerobic exercise regimen in those with more advanced disease as well as gathering preliminary data on the impact it will have on motor and nonmotor features in this cohort. In addition to the clinical outcomes, investigators are now able to capture neuronal activity with novel FDA-approved DBS technology, allowing us to non-invasively monitor real-time changes in the basal ganglia in those who have undergone DBS surgery. This study will also aim to characterize baseline neuronal activity in this cohort and monitor for changes that occur during exercise as well as determine if there is a change in baseline neuronal activity as exercise tolerance improves and with consistent, regular aerobic exercise.

ELIGIBILITY:
Inclusion criteria:

* Individuals with Parkinson's Disease
* Age >18
* H&Y stage 1-3 in the medication on and stimulation on state
* History of STN DBS
* Able to tolerate exercise from a cardiovascular, cognitive, and orthopedic perspective
* Not on beta-blockers, as we will be using heart rate-based targets
* Stable medication and stimulation for 60 days prior to baseline visit
* Access to exercise equipment

Exclusion criteria:

* Medical comorbidities that preclude safe exercise per the discretion of the principal investigator
* Regular exercisers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of study participants who complete at least 80% of the exercise sessions during the 3-month follow-up period | Following 3-month exercise regimen
  For Objective #1, feasibility of the aerobic exercise regimen will be assessed by the adherence proportion, defined as proportion of study participants who complete at least 80% of the exercise sessions during the 3-month follow-up period. Precision of the proportion estimate will be assessed by the 95% Clopper-Pearson confidence interval (CI).

SECONDARY OUTCOMES:
Change in MDS-NMS score | Following 3-month exercise regimen
  For Objective #2, the primary outcome, the change in total (Movement Disorder Society - Non-Motor Scale (MDS-NMS) score from baseline to three months. MDS-NMS is reported as a score from 0-334, with higher scores being worse. In secondary analysis we will summarize and compare the score of each individual domain between the two time points (depression, anxiety, apathy, psychosis, impulse control, cognition, orthostatic hypotension, urinary, sexual, gastrointestinal, sleep, pain, and other).
Change in number of symptoms reported | Following 3-month exercise regimen
  Proportion of subjects with each non-motor symptom (with score of at least 1). The total number of symptoms and number of symptoms within each domain will be compared using the Wilcoxon signed-rank test.
Change in LFP | Following 3-month exercise regimen
  For the exploratory objective to study changes in neuronal activity, we will use linear and non-linear mixed effects models to study the trend in the biweekly measurements of local field potentials (LFPs) parameters over time. The LFP parameters, including power, sample entropy, arrhythmicity, and asymmetry primarily in beta bands but will also explore other frequencies, will be transformed, if needed, to achieve approximate normality. Random intercepts based on patient and STN will be included in the model. In addition, changes in LFP parameters from baseline to various time points will be associated with changes in total and domain-specific MDS-NMS scores from baseline to three months using linear regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Aslam, DO, Principal Investigator — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No